CLINICAL TRIAL: NCT02369471
Title: A Double Blind, Randomized, Placebo-controlled, Two-part Study to Investigate the Pharmacokinetics, Followed by Efficacy and Safety of GWP42006 as add-on Therapy in Patients With Inadequately Controlled Focal Seizures.
Brief Title: A Study of GWP42006 in People With Focal Seizures - Part A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GWEP1330 Part A; 2014-002594-11 (EudraCT Number)
Record Dates: First submitted 2015-02-13; First posted 2015-02-24 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Epilepsy; Focal Seizures
Keywords: Cannabidivarin; CBDV; GWP42006
MeSH Terms: conditions — Epilepsy; Seizures | interventions — cannabidivarin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1a (Experimental): Subjects on inducer AEDs will administer GWP42006.
  Interventions: Drug: GWP42006
- Group 2a (Active Comparator): Subjects on inhibitor AEDs will administer GWP42006.
  Interventions: Drug: GWP42006
- Group 3a (Experimental): Subjects on AEDs that are neither inducers nor inhibitors will administer GWP42006.
  Interventions: Drug: GWP42006
- Group 1b (Placebo Comparator): Matching placebo control for Group 1a.
  Interventions: Drug: Placebo
- Group 2b (Placebo Comparator): Matching placebo control for Group 2a.
  Interventions: Drug: Placebo
- Group 3b (Placebo Comparator): Matching placebo control for Group 3a.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GWP42006
  Other Names: Cannabidivarin; CBDV
  Arms: Group 1a; Group 2a; Group 3a
Drug: Placebo
  Arms: Group 1b; Group 2b; Group 3b

SUMMARY:
To evaluate the pharmacokinetics, safety and tolerability of GWP42006 compared with placebo, in the presence of other antiepileptic drugs (AEDs).

DETAILED DESCRIPTION:
This is a double blind, randomized, placebo controlled, two-part study. Part A only will be described in this record.

Subjects who satisfy all inclusion and none of the exclusion criteria will begin a 14-day baseline observation period followed by a 14-day treatment period. Subjects will be required to attend six study visits. A follow-up phone call will take place four weeks after last dose.

Part A will enroll three groups of 10 subjects:

* Group 1 - subjects on inducer AEDs (and not on inhibitor AEDs)
* Group 2 - subjects on inhibitor AEDs (and not on inducer AEDs)
* Group 3 - subjects on AEDs that are neither inducers nor inhibitors.

In each of the three groups subjects will be randomized to receive, in a 4:1 ratio, GWP42006 400 mg twice daily or matching placebo. Pharmacokinetic (PK) profiles for GWP42006 and metabolites will be collected on the first and last day of treatment. Samples will also be collected 24h and 72h after the last day of treatment.

Subjects will be required to record a daily diary with information about their seizures, investigational medicinal product (IMP) and concomitant AED administration.

ELIGIBILITY:
For inclusion in Part A of the study patients must fulfil ALL of the following criteria:

* Male or female aged between 18 and 65 years, inclusive.
* Well-documented history of focal epilepsy, with focal seizures as the primary seizure type, compatible electroencephalogram and clinical history.
* Documented computerized tomography / magnetic resonance imaging that shows no progressive neurologic abnormality.
* Has focal seizures despite prior treatment with at least two AEDs (whether as monotherapies or in combination).
* Currently treated with one to three AEDs as follows:

  * Group 1 - subjects on inducer AEDs (and not on inhibitor AEDs)
  * Group 2 - subjects on inhibitor AEDs (and no on inducer AEDs)
  * Group 3 - subjects on AEDs that are neither inducers nor inhibitors.
* All medications or interventions for epilepsy (including ketogenic diet and any neurostimulation devices for epilepsy) must have been stable for two weeks prior to screening and the patient is willing to maintain a stable regimen throughout the study.
* Subject is willing to keep any factors expected to affect seizures stable (such as the level of alcohol consumption and smoking).

The patient may not enter Part A of the study if ANY of the following apply:

* Time of onset of epilepsy treatment is less than two years prior to enrolment.
* Episode(s) of status epilepticus during one year prior to screening.
* History of pseudo-seizures.
* Subject has clinically significant unstable medical conditions other than epilepsy.
* Subject has an illness in the four weeks prior to screening or randomization, other than epilepsy, which in the opinion of the investigator would affect seizure frequency.
* Subject has significantly impaired hepatic function at Visit 1.
* Active suicidal plan/intent in the past six months, or a history of suicide attempt in the last two years, or more than one lifetime suicide attempt.
* Subject is currently using or has in the past used recreational or medicinal cannabis, or cannabinoid based medications within the three months prior to screening and is unwilling to abstain for the duration for the study.
* Subject has taken St John's Wort in the last two weeks and/or is unwilling to abstain throughout the study.
* Subject has consumed grapefruit or grapefruit juice three days prior to randomization and/or unwilling to abstain in the three days prior to Visits A2 and A4.
* Any known or suspected hypersensitivity to cannabinoids, sesame oil or any of the excipients of the IMP(s).
* Subjects who have received an IMP within the 12 weeks prior to the screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of GWP42006 and metabolites: Cmax, Cmin, tmax, AUC(0-t), AUC(0-inf) and t1/2, in the presence of other AEDs. | Day 1 to Day 18

SECONDARY OUTCOMES:
Safety and tolerability of GWP42006 (incidence of adverse events). | Day -14 to Day 43
The plasma concentration of concomitant AEDs. | Day 1 and Day 15

CONTACTS AND LOCATIONS:
Locations (9):
- Czechia (3):
  - Havířov
  - Hradec Králové
  - Rychnov nad Kněžnou
- Barcelona, Spain
- United Kingdom (5):
  - Birmingham
  - Dundee
  - Glasgow
  - Great Yarmouth
  - Stoke-on-Trent